CLINICAL TRIAL: NCT01364428
Title: A Trial Comparing the Efficacy and Safety of Insulin Degludec 200 U/mL and Insulin Degludec 100 U/mL in Subjects With Type 2 Diabetes Mellitus (BEGIN™: COMPARE)
Brief Title: Comparison of Two Insulin Degludec Formulations in Subjects With Type 2 Diabetes Mellitus
Acronym: BEGIN™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-3923; U1111-1119-2518 (Registry Identifier: WHO)
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Results first posted 2015-11-18 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDeg 200 U/mL (Experimental)
  Interventions: Drug: insulin degludec
- IDeg 100 U/mL (Experimental)
  Interventions: Drug: insulin degludec

INTERVENTIONS:
Drug: insulin degludec — Injected subcutaneously (under the skin) once daily, in combination with unchanged pre-trial oral anti-diabetic drug (OAD) treatment.
  Dose was individually adjusted.
  Arms: IDeg 200 U/mL
Drug: insulin degludec — Injected subcutaneously (under the skin) once daily, in combination with unchanged pre-trial oral anti-diabetic drug (OAD) treatment.
  Dose was individually adjusted.
  Arms: IDeg 100 U/mL

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this trial is to compare the efficacy and safety of two different formulations of insulin degludec (IDeg) in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes (diagnosed clinically) for minimum 24 weeks prior to randomisation (visit 2)
* Current treatment with basal-only insulin (no prandial insulin) consisting of either insulin detemir once daily (OD), insulin glargine OD or neutral protamine hagedorn (NPH) insulin OD/twice daily (BID) for at least 12 weeks prior to randomisation (visit 2), in combination with stable doses of OAD(s) (metformin, insulin secretagogue (sulfonylurea or glinide), alpha-glucosidase inhibitor, pioglitazone or dipeptidyl peptidase IV (DPP-IV) inhibitor in any approved (according to label) dose or combination. Stable OAD doses are defined as unchanged doses for at least 12 weeks prior to randomisation (visit 2)
* HbA1c (glycosylated haemoglobin) between 7.0-10.0% (both inclusive) by central laboratory analysis
* Body mass index (BMI) below or equal to 45 kg/m^2
* Ability and willingness to adhere to the protocol including self-measured plasma glucose (SMPG) according to the protocol

Exclusion Criteria:

* Treatment with rosiglitazone within the last 12 weeks prior to randomisation (visit 2)
* Treatment with glucagon like peptide-1 (GLP-1) receptor agonists within the last 12 weeks prior to randomisation (visit 2)
* Recurrent severe hypoglycaemia (more than one severe hypoglycaemic event during the last 12 months) or hypoglycaemic unawareness as judged by the Investigator (trial physician)
* Previous participation in this trial. Participation is defined as randomised. Re-screening is allowed once during the recruitment period
* Known or suspected hypersensitivity to trial products or related products
* The receipt of any investigational drug within 4 weeks prior to randomisation (visit 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 373 (Actual)
Dates: Start 2011-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (43):
- United States (43):
  - Novo Nordisk Investigational Site, Huntsville, Alabama
  - Novo Nordisk Investigational Site, Goodyear, Arizona
  - Novo Nordisk Investigational Site, Mesa, Arizona
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Greenbrae, California
  - Novo Nordisk Investigational Site, Montclair, California
  - Novo Nordisk Investigational Site, National City, California
  - Novo Nordisk Investigational Site, Palm Springs, California
  - Novo Nordisk Investigational Site, Bradenton, Florida
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, Kissimmee, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, West Palm Beach, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Springfield, Illinois
  - Novo Nordisk Investigational Site, Evansville, Indiana
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, Slidell, Louisiana
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Waltham, Massachusetts
  - Novo Nordisk Investigational Site, Detroit, Michigan
  - Novo Nordisk Investigational Site, Jefferson City, Missouri
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Lawrenceville, New Jersey
  - Novo Nordisk Investigational Site, Toms River, New Jersey
  - Novo Nordisk Investigational Site, Staten Island, New York
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Canton, Ohio
  - Novo Nordisk Investigational Site, Franklin, Ohio
  - Novo Nordisk Investigational Site, Melrose Park, Pennsylvania
  - Novo Nordisk Investigational Site, Brentwood, Tennessee
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Hurst, Texas
  - Novo Nordisk Investigational Site, Irving, Texas
  - Novo Nordisk Investigational Site, Round Rock, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Olympia, Washington
  - Novo Nordisk Investigational Site, Renton, Washington

REFERENCES:
- [Result] Bode BW, Chaykin LB, Sussman AM, Warren ML, Niemeyer M, Rabol R, Rodbard HW. Efficacy and Safety of Insulin Degludec 200 U/mL and Insulin Degludec 100 U/mL in Patients with Type 2 Diabetes (Begin: Compare). Endocr Pract. 2014 Aug;20(8):785-91. doi: 10.4158/EP13411.OR. PMID 24518180
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 44 sites within United States of America.
Pre-assignment Details: Subjects who were treated with basal insulin in combination with unchanged dosing of oral antidiabetic drug treatment (e.g. metformin, pioglitazone or DPP-IV inhibitor) in any approved dose or combination at unchanged dosing for at least 12 weeks prior to randomisation in a 1:1 manner to IDeg 200 U/mL or IDeg.
Groups:
- IDeg 200 U/mL: Insulin degludec 200 U/mL (IDeg 200 U/mL) in a 3 mL prefilled pen PDS290 was given subcutaneously once daily in combination with pre-trial oral antidiabetic drug treatment(metformin, insulin secretagogue [sulfonylurea or glinide], alpha-glucosidase inhibitor, pioglitazone or DPP-IV inhibitor). IDeg 200 U/mL was administered at any time of the day but preferably at the same time each day.
- IDeg: Insulin degludec 100 U/mL (IDeg) in a 3 mL prefilled pen PDS290 was given subcutaneously once daily in combination with pre-trial oral antidiabetic drug treatment (metformin, insulin secretagogue [sulfonylurea or glinide], alpha-glucosidase inhibitor, pioglitazone or DPP-IV inhibitor). IDeg was administered at any time of the day but preferably at the same time each day.
Period: Overall Study
Arm/Group | IDeg 200 U/mL | IDeg
Started | 186 | 187
Exposed | 184 (Two subjects were randomised in error and withdrew prior to exposure to drug) | 187
Completed | 166 | 172
Not Completed | 20 | 15
Not completed — Adverse Event | 1 | 2
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal Criteria | 14 | 10
Not completed — Other | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDeg 200 U/mL | IDeg | Total
Number analyzed (Participants) | 186 | 187 | 373
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (10.0) | 60.3 (10.2) | 59.8 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 70 | 168
  Male | 88 | 117 | 205
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.1 (0.9) | 8.2 (0.9) | 8.2 (0.9)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 8.3 (3.0) | 8.3 (3.4) | 8.3 (3.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Change from baseline in HbA1c after 22 weeks of treatment
Time Frame: Week 0, Week 22
Population: The full analysis set (FAS) included all randomised subjects and missing data was imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDeg 200 U/mL | IDeg
Number analyzed (Participants) | 186 | 187
percentage of glycosylated haemoglobin | -0.79 (0.89) | -0.70 (0.90)

2. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change from baseline in FPG after 22 weeks of treatment.
Time Frame: Week 0, Week 22
Population: The full analysis set (FAS) included all randomised subjects and missing data was imputed using last observation carried forward (LOCF). For 5 subjects baseline values were missing.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg 200 U/mL | IDeg
Number analyzed (Participants) | 182 | 186
mmol/L | -2.26 (3.07) | -2.40 (3.42)

3. Secondary Outcome: Rate of Treatment Emergent Adverse Events (AEs)
Description: Corresponds to rate of AEs per 100 patient years of exposure. Severity assessed by investigator. Mild: no or transient symptoms, no interference with subject's daily activities. Moderate: marked symptoms, moderate interference with subject's daily activities. Severe: considerable interference with subject's daily activities, unacceptable. Serious AE: AE that at any dose results in any of the following: death, a life-threatening experience, in-subject hospitalization/prolongation of existing hospitalisation, persistent/significant disability/incapacity/congenital anomaly/birth defect.
Time Frame: Week 0 to Week 22 + 7 days follow up
Population: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: Events/100 years of patient exposure
Arm/Group | IDeg 200 U/mL | IDeg
Number analyzed (Participants) | 184 | 187
Events/100 years of patient exposure
  Adverse events (AEs) | 416 | 300
  Serious AEs | 20 | 16
  Severe AEs | 27 | 21
  Moderate AEs | 130 | 107
  Mild AEs | 259 | 172
  Fatal AEs | 0 | 0

4. Secondary Outcome: Rate of Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes were defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes were defined as able to treat her/himself and plasma glucose below 3.1 mmol/L.
Time Frame: Week 0 to Week 22 + 7 days follow up
Population: as for outcome 3
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDeg 200 U/mL | IDeg
Number analyzed (Participants) | 184 | 187
Episodes/100 years of patient exposure | 517 | 566

5. Secondary Outcome: Rate of Nocturnal Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes were defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes were defined as able to treat her/himself and plasma glucose below 3.1 mmol/L. Nocturnal hypoglycaemic episodes were defined as occurring between 00:01 and 05:59 a.m.
Time Frame: Week 0 to Week 22 + 7 days follow up
Population: as for outcome 3
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDeg 200 U/mL | IDeg
Number analyzed (Participants) | 184 | 187
Episodes/100 years of patient exposure | 127 | 170

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time frame of 22 weeks + 7 days follow up.
Description: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator.
Arm/Group | IDeg 200 U/mL | IDeg
Serious Adverse Events (participants affected / at risk) | 9/184 | 11/187
Other Adverse Events (participants affected / at risk) | 45/184 | 26/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg 200 U/mL (N=184) | IDeg (N=187)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tongue neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Drug abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg 200 U/mL (N=184) | IDeg (N=187)
Diarrhoea (Gastrointestinal disorders) | 17 (20) | 4 (4)
Nasopharyngitis (Infections and infestations) | 18 (19) | 12 (14)
Upper respiratory tract infection (Infections and infestations) | 15 (17) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.